CLINICAL TRIAL: NCT07396844
Title: A Single Dose, Randomized, Open-label, Two-way Crossover Food-effect Bioavailbility Study of Fixed Dose Combination of Gemigliptin/Dapagliflozin/Metformin 50/10/1000 mg Sustained Release Tablets Under Fasting and Fed Conditions in Healthy Volunteers
Brief Title: The Food Effect on Pharmacokinetics of Fixed Dose Combination of Gemigliptin/Dapagliflozin/Metformin in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-GMCL002
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Healthy; Fasting; Fed
MeSH Terms: conditions — Fasting; Lecithin Cholesterol Acyltransferase Deficiency | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 : Period 1 (Fasting) - Period 2 (Fed)
  Interventions: Drug: Fixed-dose combination of gemigliptin/dapagliflozin/metformin 50/10/1000 mg
- Group 2 (Experimental): Group 2 : Period 1 (Fed) - Period 2 (Fasting)
  Interventions: Drug: Fixed-dose combination of gemigliptin/dapagliflozin/metformin 50/10/1000 mg

INTERVENTIONS:
Drug: Fixed-dose combination of gemigliptin/dapagliflozin/metformin 50/10/1000 mg — All participants will receive a single tablet of the study drug (a fixed-dose combination of gemigliptin/dapagliflozin/metformin 50/10/1000 mg) under either fasting or fed conditions.

SUMMARY:
This is a single dose, randomized, open-label, two-way crossover study to investigate the food-effect bioavailability of the fixed-dose combination of Gemigliptin/Dapagliflozin/Metformin 50/10/1000 mg in healthy volunteers under fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Thai male and female subjects between the ages of 18 to 55 years.
2. Body mass index between 18.5 to 30.0 kg/m2.
3. Normal laboratory values, including vital signs and physical examination, for all parameters in clinical laboratory tests at screening.
4. Non-pregnant woman and not currently breast feeding.
5. Female subjects abstain from either hormonal method of contraception or hormone replacement therapy.
6. Male subjects who are willing or able to use effective contraceptive.
7. Have voluntarily given written informed consent by the subject prior to participating in this study.

Exclusion Criteria:

1. History of allergic reaction or hypersensitivity to gemigliptin or dapagliflozin or metformin.
2. History of evidence of clinically significant renal, hepatic, gastrointestinal, hematological, endocrine, pulmonary or respiratory, cardiovascular, neurologic, allergic disease, or any significant ongoing chronic medical illness.
3. History of evidence of diabetic ketoacidosis.
4. History of evidence of genital infections, urinary tract infections within 14 days prior to check-in.
5. Have a eGFR (CKD-EPI) < 60 mL/min/1.73 m2.
6. History or evidence of alcoholism or harmful use of alcohol within 2 years prior to screening.
7. Participated in other clinical trial within 90 days prior to check-in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin. | 17 times up to 72 hours after IP administration
  Primary PK Parameters: Area under the plasma concentration versus time curve (AUClast) of Gemigliptin, Dapagliflozin, and Metformin
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin. | 17 times up to 72 hours after IP administration
  Primary PK Parameters: Area Under the Curve to Infinity (AUCinf) of Gemigliptin, Dapagliflozin, and Metformin
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin. | 17 times up to 72 hours after IP administration
  Peak Plasma Concentration (Cmax) of Gemigliptin, Dapagliflozin, and Metformin

SECONDARY OUTCOMES:
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin. | 17 times up to 72 hours after IP administration
  Secondary PK Parameters: Time to Maximum(Tmax) Concentration of gemigliptin, dapagliflozin, and metformin
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin. | 17 times up to 72 hours after IP administration
  Secondary PK Parameters: Half-life(t1/2) of gemigliptin, dapagliflozin, and metformin

OTHER OUTCOMES:
Assessment - Safety (Adverse events) | Up to Day 4 (72 hours)
  A list of all adverse events for each treatment group and for all participants with seriousness, severity, relationship with investigational product. A number of participant with adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Porranee Puranajoti, Principal Investigator — International Bio Service Co., Ltd.
Locations (1):
- Siriraj Hospital, Nakhon Phanom, Thailand

IPD SHARING:
Plan to Share IPD: No